CLINICAL TRIAL: NCT03233035
Title: Intranasal Ketamine for Treatment of Acute Pain in the Emergency Department : A Randomized Controlled Trial
Brief Title: Low Dose Ketamine Intra Nasal Traumatology
Acronym: Ket
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ket-Int-Nas-TR
Record Dates: First submitted 2017-05-14; First posted 2017-07-28 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Trauma
Keywords: Ketamine-Intranasal-Acute pain-Emergency departement
MeSH Terms: conditions — Wounds and Injuries | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double Blind Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Ketamine versus placebo as a double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo group (Placebo Comparator): Intranasal placebo pulverisation
  Interventions: Drug: Placebo
- Ketamine group (Active Comparator): Intranasal ketamine pulverisation
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 25mg of ketamine in 0.5 ml of serum saline in one pulverisation per nostril is received
  Arms: Ketamine group
Drug: Placebo — 0.5 mL of normal saline solution as a placebo in one pulverisation per nostril
  Other Names: normal saline solution
  Arms: placebo group

SUMMARY:
To evaluate the efficacy and safety of early administration of low-dose intranasal ketamine analgesic agents in patients with moderate to severe pain in the ED in reducing the need for opioid or non opioids analgesic agents.

DETAILED DESCRIPTION:
Intranasal ketamine for treatment of acute pain in the emergency department : A randomized controlled trial

Introduction :

Pain is the most common complaint for emergency department (ED) visits [1].The provision of adequate, safe, and timely analgesia is a core component of patient care in the emergency department (ED). Ketamine is a noncompetitive Nmethyl- D-aspartate and glutamate receptor antagonist that decreases central sensitization, "wind-up" phenomena, and pain memory [2,3].

At subdissociative doses (0.1 to 0.6 mg/kg; most commonly 0.3 mg/kg) maintains potent analgesic and amnestic effects that are accompanied by preservation of protective airway reflexes, spontaneous respiration, and cardiopulmonary stability [4-6].

Intranasal route ….

Objective of the study :

To evaluate the efficacy and safety of early administration of low-dose intranasal ketamine analgesic agents in patients with moderate to severe pain in the ED in reducing the need for opioid or class III analgesic agents.

Materials and Methods :

Study design :

It is a ramdomized, prospective, double blind, controlled, multicentric trial. The study is registered with clinical.tria.gov (…….).

Study Setting and Selection of Participants :

The trial is conducted in three community teaching hospitals :

* Emergency department, fattouma bourguiba university hospital, monastir, tunisia
* Emergency department, sahloul university hospital, sousse, tunisia
* Emergency department, farhat hached university hospital, sousse, tunisia

ED principal investigators maintain the randomization list, which is generated before the start of the study, prepare the medication, and deliver it to the treating physician in a blinded manner.

Inclusion criteria :

The study includes patients aged 18 to 80 years who presented to the ED with acute limb trauma pain with a visual analogue scale (VAS) of 5 or more on a standard 11- point (0 to 10). An informed consent is necessary.

Exclusion criteria :

* Pregnancy,
* Breast-feeding,
* Altered mental status,
* Allergy to ketamine or morphine or
* Weight less than 46 kg or greater than 115 kg,
* Unstable vital signs (systolic blood pressure <90 or >180 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min),
* Medical history of acute head or eye injury, seizure, intracranial hypertension, chronic pain, severre renal or hepatic insufficiency,
* Alcohol or drug abuse,
* Psychiatric illness,
* Recent (4 hours before) analgesic agent use.

Protocol :

In the triage area, each patient having the inclusion criteria receives 25mg of ketamine in 0.5 ml of serum saline in one pulverisation per nostril or 0.5 mL of normal saline solution in one pulverisation per nostril as a placebo according to the predetermined randomization list. None of the treating physician or nurses is aware about the medication received. In all patients included, the investigators collect vital signs ; demographic and clinical data.

Study investigators record VAS, and adverse effects at 15, 30, 60, 90, and 120 minutes.

At 30 minutes, if patients report a pain numeric rating scale score of 5 or greater and request additional pain relief, titrated morphine is administered as a rescue analgesic with a dose of 0.1 mg/Kg repeated every 3 to 5 minutes if the pain numeric rating scale score is still greater or equal to 3.

All data recorded on data collection sheets, including sex, demographics, medical history, and vital signs, were entered into SPSS (version 20.0; IBM Corp) by the research manager.

Patients's informed consent is obtained. The ethic commitee of our institution approved the study.

Endpoints :

Primary endpoints :

- Need for rescue opioids during ED stay

Secondary endpoints :

* requirement of non-opioids analgesic agents.
* percentage of patients discharged from the ED with VAS <30.
* Safety : adverse events

ELIGIBILITY:
Inclusion Criteria:

* The study includes patients aged 18 to 80 years who presented to the ED with acute limb trauma pain with a visual analgesic scale (VAS) of 5 or more on a standard 11- point (0 to 10). An informed consent is necessary.

Exclusion Criteria:

* - Pregnancy,
* Breast-feeding,
* Altered mental status,
* Allergy to ketamine or morphine or
* Weight less than 46 kg or greater than 115 kg,
* Unstable vital signs (systolic blood pressure <90 or >180 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min),
* Medical history of acute head or eye injury, seizure, intracranial hypertension, chronic pain, severre renal or hepatic insufficiency,
* Alcohol or drug abuse,
* Psychiatric illness,
* Recent (4 hours before) analgesic agent use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients who need rescue opiods in the two groups | 30 minutes
  the need for rescue opioids during ED stay

SECONDARY OUTCOMES:
Intolerance to treatement and adverse events | 30 minutes and at 120 minutes
  Noticing any sign of intolerance due to treatement : Dizziness , Vomiting..
Percentage of patients with VAS <30 mm at discharge | 120 minutes
  percentage of patients discharged from the ED with VAS <30.
Number and percentage of patients who required non opiods analgesics | 30 minutes
  Requirement of non-opioids analgesic agents

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — university Hospital of Monastir
Locations (2):
- Tunisia (2):
  - Nouira Samir, Monastir, Emergency Department Monastir, Tunisia 5000
  - Emergency department of university hospital Fattouma Bourguiba of Monastir, Monastir

IPD SHARING:
Plan to Share IPD: No